CLINICAL TRIAL: NCT06435949
Title: Effect of Propofol in Combination With Oxycodone on Anxiety State in Painless Abortion - A Multicenter Randomized Controlled Trial
Brief Title: Effect of Oxycodone on Anxiety State in Painless Abortion
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: RJH-Anesth-HZH001
Record Dates: First submitted 2024-03-31; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-03

CONDITIONS: Abortion Complication
MeSH Terms: interventions — Fentanyl; Oxycodone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group Fentanyl (Experimental): intravenous anesthesia with propofol with fentanyl
  Interventions: Drug: Fentanyl (as Citrate)
- group Oxycodone (Experimental): intravenous anesthesia with propofol with oxycodone
  Interventions: Drug: Fentanyl (as Citrate)

INTERVENTIONS:
Drug: Fentanyl (as Citrate) — intravenous anesthesia with propofol with fentanyl (group Fentanyl) and propofol with oxycodone (group Oxycodone)
  Other Names: Oxycodone

SUMMARY:
In this study, 300 patients who underwent painless abortion in Ruijin Hospital and sub-central hospitals were selected through a multi-center randomized controlled study, and 300 patients who underwent painless abortion in Ruijin Hospital and each sub-center hospital were divided into intravenous anesthesia with propofol with fentanyl (group F) and propofol with oxycodone (group O) by stratified group randomization method 1:1. The difference between the postoperative anxiety scores and depression scores of the two groups was observed, and the postoperative anxiety, depression and numerical pain scores were recorded. Finally, the relevant data were statistically analyzed and conclusions were drawn.

DETAILED DESCRIPTION:
This study is a multicenter, randomized controlled clinical study. A total of 300 patients who underwent elective painless abortion surgery in Ruijin Hospital and other sub-central hospitals were enrolled, and they were randomly divided into 1:1 patients who received intravenous anesthesia with propofol with fentanyl (group F) and propofol with oxycodone (group O). The scores of anxiety, depression and postoperative numerical rating scale (NRS) before and after surgery were observed, and the levels of serum stress response factors and inflammatory cytokines were monitored. The effects of oxycodone on anxiety, depression and postoperative acute pain in patients with painless abortion were investigated.

1. Main observation indicators:

   The difference between the post-operative anxiety score and the preoperative anxiety score
2. Secondary Observational Indicators:

   * Post-operative anxiety score
   * The difference between the post-operative depression score and the preoperative depression score
   * Post-operative depression score
   * Pain assessment after surgical recovery (NRS)
   * Laboratory tests
   * Patient and family satisfaction with postoperative analgesic treatment

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45 years old
* Gestational age 6-12 weeks
* American Society of Anesthesiologists （ASA） Grading I-II
* Fluent communicator and able to complete self-rating scales on her own
* Voluntarily participate and sign the informed consent form

Exclusion Criteria:

* Patients who are allergic to anesthetic drugs such as propofol, oxycodone, fentanyl, etc., or who have had other anesthetic adverse events
* Patients with anxiety or depression
* Presence of organic mental disorders, mental retardation
* Severe acute and chronic infection, severe heart, liver and kidney insufficiency
* Patients with complications or bleeding > 50ml during surgery

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
anxiety scores | 20-30 minutes postoperative
  postoperative anxiety scores

SECONDARY OUTCOMES:
depression scores | 20-30 minutes postoperative
  postoperative depression scores

IPD SHARING:
Plan to Share IPD: No